CLINICAL TRIAL: NCT02368873
Title: Prospective, Randomized Study on the Use of a Intraperitoneal Onlay Mesh for Prevention of Parastomal Hernia of Permanent Colostomy
Brief Title: the Use of a IPOM Mesh for Prevention of Parastomal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Vaasa Central Hospital, Vaasa, Finland (Other); Päijänne Tavastia Central Hospital (Other); Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Tero Rautio, M.D., Ph.D., Consultant colorectal surgeon, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109/2009
Record Dates: First submitted 2014-12-19; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Parastomal Hernia
Keywords: prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Patients with IPOM Dynamesh mesh around the straight permanent colostomy.
  Interventions: Procedure: Application of IPOM mesh
- Control group (No Intervention): Patients with the straight permanent colostomy without a mesh.

INTERVENTIONS:
Procedure: Application of IPOM mesh
  Other Names: Dual-component mesh (Dynamesh IPOM, FEG Textiltechnik mbH, Aachen, Germany)
  Arms: Intervention group

SUMMARY:
Study is a prospective, multicenter, randomized trial evaluating whether prophylactic laparoscopic placement of a dual-component IPOM mesh around a colostomy may prevent parastomal hernia compared with conventional colostomy after abdominoperineal resection. Eligible subjects will be recruited prospectively from five Finnish Hospitals (Oulu University Hospital,Vaasa Central Hospital, Helsinki University Hospital, Lahti Central Hospital, Jyväskylä Central Hospital). Patients were considered eligible for this study if undergoing laparoscopic abdominoperineal resection for rectal adenocarcinoma. Patients are randomized to prophylactic preperitoneal placement of a dual-component mesh (Dynamesh IPOM) around permanent colostomy or to conventional permanent colostomy. Estimating a parastomal hernia rate of 50%, a sample size of 26 patients per each study group is projected to provide 90% power (1-beta) with a alpha 0.05 (2-beta) to detect a 40% reduction in risk for parastomal hernia at 1-year. Since we expect a dropout rate of 20%, 37 patients per study group will be included in this study.

All abdominoperineal resections are performed using laparosopic technique. At the and of the abdominal laparoscopic phase the straight permanent end colostomy is performed. In the intervention group the 10 x 10 cm Dynamesh IPOM mesh is cut in the middle according to volume of the bowel. Stapled bowel end is then pulled through the crosswise opened mesh, which is pushed to the abdomen and fixed to the peritoneum.

Follow-up visits are scheduled at 1-, 3- and 12-month after surgery. Patients are evaluated for their clinical status and C-reactive protein, leukocytes and hemoglobin are assessed at each control visit. Computed tomography (CT) scan with and without Valsalva maneuver is performed 12 months after surgery for radiological evaluation of possible parastomal hernia.

The primary end-point of this study is the incidence of clinically and radiologically detected parastomal hernias, and their extent 12 months after surgery. The secondary outcome end-points were colostomy-related morbidity such as stomal stenosis, necrosis and/or wound infection.The extent of parastomal hernia was graded at CT according to the Hernia Society criteria.

Statistical analysis is performed using a SPSS statistical software. Continuous variables are reported as the mean and standard deviation, whereas nominal variables are reported as counts and proportions. Univariate analysis is performed with the Mann-Whitney U test and Fisher's exact test. P-values < 0.05 are considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic abdominoperineal resection for rectal adenocarsinoma

Exclusion Criteria:

* Patients who can not give their consent to participate in the study
* Patients in poor general conditions (American Society of Anaesthesiologists classes 4-5)
* Patients with incurable cancer or another rectal malignancy than adenocarcinoma
* Patients with any abdominal infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of parastomal hernia | One year

SECONDARY OUTCOMES:
Number of colostomy-related complications | One year

REFERENCES:
- [Derived] Makarainen-Uhlback EJ, Klintrup KHB, Vierimaa MT, Carpelan-Holmstrom MA, Kossi JAO, Kairaluoma MV, Ohtonen PP, Tahvonen PR, Rautio TT. Prospective, Randomized Study on the Use of Prosthetic Mesh to Prevent a Parastomal Hernia in a Permanent Colostomy: Results of a Long-term Follow-up. Dis Colon Rectum. 2020 May;63(5):678-684. doi: 10.1097/DCR.0000000000001599. PMID 32032196